CLINICAL TRIAL: NCT06442709
Title: Combined Anti-IL6R and Anticoagulation Therapy Improves Prognosis in Patients With Advanced Nasopharyngeal Carcinoma
Brief Title: Combined Anti-IL6R and Anticoagulation Therapy in Advanced NPC Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-K015
Record Dates: First submitted 2024-04-25; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-03

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: nasopharyngeal narcinoma; metastasis; extracellular vesicles; organ-organ crosstalk
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Neoplasm Metastasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined Anti-IL6R and Anticoagulation Therapy in Advanced NPC Patients (Experimental): Tocilizumab, an IL6R inhibitor, injected once a month at a dose of 4mg/kg in advanced NPC patients.
  Asprin，an anticoagulant, taken orally once daily at a dose of 100mg in advanced NPC patients.
  Interventions: Drug: Tocilizumab Asprin
- Receive placebo in Advanced NPC Patients (Placebo Comparator): Placebo replaces tocilizumab and asprin in advanced NPC patients.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tocilizumab Asprin — Tocilizumab alone, Asprin alone, Tocilizumab combined with Asprin. Tocilizumab, an IL6R inhibitor, injected once a month at a dose of 4mg/kg in advanced NPC patients.
  Asprin，an anticoagulant, taken orally once daily at a dose of 100mg in advanced NPC patients.
  Arms: Combined Anti-IL6R and Anticoagulation Therapy in Advanced NPC Patients
Other: Placebo — Placebo replaces tocilizumab and asprin in advanced NPC patients.
  Arms: Receive placebo in Advanced NPC Patients

SUMMARY:
The investigators have demonstrated the crucial role of the liver-lung axis in the distant metastasis of NPC. Furthermore, the investigators have identified a potential therapeutic approach to improve outcomes in NPC patients by identifying those most suitable for anticoagulant therapy. Further, the combination of anticoagulant therapy and anti-IL6R therapy has shown promising results in enhancing the prognosis of NPC patients. These findings highlight the significance of targeting the liver-lung axis and utilizing personalized treatment strategies for NPC.

DETAILED DESCRIPTION:
Distant metastasis accounts for nasopharyngeal carcinoma (NPC)-related mortalities. Recently, extracellular vesicles (EVs) have been widely explored as key mediators of bidirectional tumor-host cell interactions by mediating pre-metastatic niche (PMN) formation. However, considering the complexity of the human body, multiple organ studies of tumor metastasis remain poorly understood. Here, the investigators have demonstrated the crucial role of the liver-lung axis in the distant metastasis of NPC. The investigators demonstrated mechanistically that hepatocellular derived EVs can be specifically taken up by the lung to form a hypercoagulable pre-metastatic microenvironment associated with IL6.Furthermore, the investigators have identified a potential therapeutic approach to improve outcomes in NPC patients by identifying those most suitable for anticoagulant therapy. Further, the combination of anticoagulant therapy and anti-IL6R therapy has shown promising results in enhancing the prognosis of NPC patients. These findings highlight the significance of targeting the liver-lung axis and utilizing personalized treatment strategies for NPC.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of NPC with distant metastasis
* Must be able to swallow tablets

Exclusion Criteria:

* Liver disease
* Blood disease
* Long-term use of anticoagulants

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Tumor progression and metastasis | Five to Ten years
  After the patients are diagnosed and treated, CT scans is used semi-annually to determine the progression and metastasis of tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Bo You, Doctor, Principal Investigator — Department of Otorhinolaryngology-Head and Neck Surgery, Affiliated Hospital of Nantong University
Locations (1):
- Bo You, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, statistical analysis plan, informed consent form, clinical study report, and analytic code will be shared to other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Two years after this clinical trial finished.
Access Criteria: Researchers must clearly state the purpose of their study and ensure it aligns with the scientific objectives of the data sharing initiative. A detailed research plan, including research design, data analysis methods, and expected results, should be provided to ensure the data is used in a reasonable and effective manner. Additionally, researchers must outline data security and privacy protection measures to ensure the safe storage, transmission, and use of the data in compliance with relevant regulations and policies.